CLINICAL TRIAL: NCT02242721
Title: Drugmonitoring of Antiinfective Drugs in Patients Receiving Continous Veno-venous Hemodiafiltration
Brief Title: Drugmonitoring of Antiinfective Drugs in Patients Receiving Continous Veno-venous Hemodiafiltration (ABx-CVVHDF)
Status: Withdrawn | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte and Campus Virchow - Klinikum, Charite University, Berlin, Germany
Other Study IDs: ABx-CVVHDF
Record Dates: First submitted 2014-09-08; First posted 2014-09-17 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Need for Renal Replacement Therapy and Anti-infective Therapy Due to Severe Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and Dialysate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intensive care unit patients needing renal replacement therapy: Male and female patients in the intensive care unit (ICU), needing renal replacement therapy due to renal dysfunction and are treated with antiinfective drugs.

SUMMARY:
Approximately 300 patients have to be enrolled in the study. They are followed up until the end of ICU stay. Usually in clinical routine, patients suspected to have infection and simultaneously renal dysfunction making CVVHDF necessary. After enrolment blood and dialysate specimens are drawn and sent for analysis on specific time points. The analysis results are sent back to the study team at the Charité - Universitätsmedizin Berlin and enable them to optimize antiinfectiva treatment of the study patients.

Data are used to test calculation tools and modify them if necessary.

DETAILED DESCRIPTION:
Little data exist whether desired and necessary blood levels of antiinfective drugs are reached during renal replacement therapy. Drug producing companies are not able to come forward with appropriate dosing recommendation in patients needing renal replacement therapy.

To achieve our study goal we plan:

1. To measure serum-concentrations of antiinfective drugs applied to the patients
2. To measure concentrations of antiinfective drugs in hemofiltration fluids.
3. To compare the actual measured concentrations with concentration predicted in known calculation tools.
4. To modify these calculation tools if necessary for better prediction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age ≥ 18 years
* Patients in the intensive care unit (ICU), needing renal replacement therapy due to renal dysfunction and are treated with antiinfective drugs

Exclusion Criteria:

* Pregnancy and lactation period.
* Participation in a clinical intervention study
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* The informed consent of the patient or the subject's legally acceptable representative can´t be obtained in time
* Patient has a power of attorney or patient's provision, where he/she refuses participation in any clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical ill patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Antibiotic clearance (l/h) | Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 5 days

SECONDARY OUTCOMES:
28-day mortality | The 28-days mortality will be assessed on the 28th study day

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Pharmacy, Kliniken Landkreis Heidenheim gGmbH, Heidenheim, Heidenheim
  - Medical Department, Division of Nephrology, Campus Charité Mitte, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin